CLINICAL TRIAL: NCT01608061
Title: A Twelve Month Double-blind Randomized Controlled Feasibility Study to Evaluate the Safety, Efficacy and Tolerability of Deep Brain Stimulation of the Fornix (DBS-f) in Patients With Mild Probable Alzheimer's Disease
Brief Title: ADvance DBS-f in Patients With Mild Probable Alzheimer's Disease
Acronym: ADvance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Functional Neuromodulation Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FNMI-001
Record Dates: First submitted 2012-05-21; First posted 2012-05-30 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer Disease
Keywords: Mild probable Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBS-f on (Experimental): DBS-f on
  Interventions: Device: DBS-f on
- DBS-f off (Sham Comparator): DBS-f off
  Interventions: Device: DBS-f off

INTERVENTIONS:
Device: DBS-f on — deep brain stimulation of the fornix
  Other Names: DBS-f system includes:; *Medtronic Activa PC Model 37601 Implantable Neurostimulator (INS); *Medtronic Model 3387 DBS Lead; *Medtronic Model 37085 DBS Extension Kit; *Medtronic Model 3708660 DBS Extension Kit
  Arms: DBS-f on
Device: DBS-f off — deep brain stimulation of the fornix turned off
  Other Names: DBS-f system includes:; *Medtronic Activa PC Model 37601 Implantable Neurostimulator (INS); *Medtronic Model 3387 DBS Lead; *Medtronic Model 37085 DBS Extension Kit; *Medtronic Model 3708660 DBS Extension Kit
  Arms: DBS-f off

SUMMARY:
The primary objective of this feasibility study is to evaluate the safety of DBS-f in patients with mild Alzheimer's disease by assessing all device and/or therapy related adverse events. The secondary objective is to preliminarily estimate the treatment effect size on the outcomes of interest at 12 months post-randomization. The objectives do not involve formal tests of hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. 45-85 years of age (inclusive)
2. Probable Alzheimer's disease according to the National Institute of Aging Alzheimer's disease Association criteria.
3. Must meet certain criteria on cognitive and behavioral rating scales
4. If female, subjects who are post-menopausal or surgically sterile or willing to use birth control methods for the duration of the study.
5. An available caregiver willing to participate.
6. Subject is living at home and likely to remain at home for the study duration.
7. The subject is currently taking a stable dose of cholinesterase inhibitor (AChEI) medication for at least 60 days

Exclusion Criteria:

1. Must meet certain criteria on cognitive and behavioral rating scales
2. Current major psychiatric disorder such as schizophrenia, bipolar disorder or major depressive disorder based on psychiatric consult at screening visit
3. History of head trauma in the 2 years prior to signing the consent to participate in the study
4. History of brain tumor, subdural hematoma, or other clinically significant (in the judgment of the investigator) space-occupying lesion on CT or MRI
5. Active psychiatric disorder
6. Mental retardation
7. Current alcohol or substance abuse as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)
8. Contraindications for PET scanning (e.g., insulin dependent diabetes)
9. Contraindications for MRI scanning, including implanted metallic devices (e.g. non-MRI-safe cardiac pacemaker or neurostimulator; some artificial joints metal pins; surgical clips; or other implanted metal parts), or claustrophobia or discomfort in confined spaces.
10. Abnormal lab results that, in the opinion of the investigator and/or enrollment review committee, would preclude participation in the study.
11. Abnormal cardiovascular or neurovascular disorder that, in the opinion of the investigator and/or enrollment review committee, would preclude participation in the study.
12. Unstable doses of any medication prescribed for the treatment of memory loss or Alzheimer's disease.
13. Currently prescribed any non-AD medications that, in the opinion of the investigator and/or enrollment review committee, would preclude participation in the study.
14. Is unable or unwilling to comply with protocol follow-up requirements.
15. Has a life expectancy of < 1 year.
16. Is actively enrolled in another concurrent clinical trial.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lozano, MD, PhD, Principal Investigator — University Health Network, Toronto; Constantine G Lyketsos, MD, MHS, DFAPA, FAPM, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (6):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Research Institute at Sun City, Sun City, Arizona
  - University of Florida at Gainesville, Gainesville, Florida
  - Johns Hopkins Bayview, Baltimore, Maryland
  - Hospital of the University of Pennsylvania: Penn Memory Clinic, Philadelphia, Pennsylvania
  - Brown University, Providence, Rhode Island
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lozano AM, Fosdick L, Chakravarty MM, Leoutsakos JM, Munro C, Oh E, Drake KE, Lyman CH, Rosenberg PB, Anderson WS, Tang-Wai DF, Pendergrass JC, Salloway S, Asaad WF, Ponce FA, Burke A, Sabbagh M, Wolk DA, Baltuch G, Okun MS, Foote KD, McAndrews MP, Giacobbe P, Targum SD, Lyketsos CG, Smith GS. A Phase II Study of Fornix Deep Brain Stimulation in Mild Alzheimer's Disease. J Alzheimers Dis. 2016 Sep 6;54(2):777-87. doi: 10.3233/JAD-160017. PMID 27567810
- [Derived] Ponce FA, Asaad WF, Foote KD, Anderson WS, Rees Cosgrove G, Baltuch GH, Beasley K, Reymers DE, Oh ES, Targum SD, Smith GS, Lyketsos CG, Lozano AM; ADvance Research Group. Bilateral deep brain stimulation of the fornix for Alzheimer's disease: surgical safety in the ADvance trial. J Neurosurg. 2016 Jul;125(1):75-84. doi: 10.3171/2015.6.JNS15716. Epub 2015 Dec 18. PMID 26684775
- See also: Study Informational Website — http://www.advancestudy4ad.com

RESULTS

PARTICIPANT FLOW:
Period: Blinded Period
Arm/Group | DBS-f on | DBS-f Off
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Long Term Follow-Up
Arm/Group | DBS-f on | DBS-f Off
Started | 21 | 21
Completed | 14 | 16
Not Completed | 7 | 5
Period: Extension Period
Arm/Group | DBS-f on | DBS-f Off
Started | 14 | 16
Completed | 14 | 14
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DBS-f on | DBS-f Off | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Median (Full Range); unit: years] | 68.1 [51.1 to 79.7] | 71.3 [48.0 to 78.0] | 69.9 [48.0 to 79.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
ADAS-Cog 11 [Median (Full Range); unit: units on a scale] — Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog 11). The cognitive subscale (ADAS-Cog) includes 11 tasks that include both subject-completed tests and observer-based assessments.Together these tasks assess the cognitive domains of memory, language, and praxis. Single scale from 0 to 70 where a higher score indicates more advanced disease.
  units on a scale | 17 [13 to 22] | 17 [12 to 21] | 17 [12 to 22]
CDR [Number; unit: Participants] — Clinical Dementia Rating scale (CDR). The CDR is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. The necessary information to make each rating is obtained through a semi-structured interview of the patient and a reliable informant or collateral source (e.g., family member). Range is 0 to 3 with a higher score indicating more advanced disease.
  Participants
    0.5 | 13 | 15 | 28
    1.0 | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Acute Safety
Description: Acute safety will be assessed by estimating the rate of serious device (pulse generator or lead) or procedure related adverse events from the date of implant through the date of randomization, plus serious procedure related events through 30 days post-implant. All subjects undergoing an implant procedure will be included in these rate estimates. The rate and 95% confidence interval will be presented. Analysis is of a timepoint prior to randomization and thus all subjects are analyzed together.
Time Frame: 30 days post implant
Population: All implanted subjects are used in this analysis. This analysis is of the entire population prior to randomization and thus cannot be analyzed per arm.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- All Implanted Subject: All implanted subjects are included in this group.
Arm/Group | All Implanted Subject
Number analyzed (Participants) | 42
participants | 2 [0.6 to 16.2]

2. Primary Outcome: Long Term Safety. Not Based on Formal Hypotheses.
Description: Long-term safety will be assessed by the rate of serious device or therapy related adverse events from the date of randomization through the date of the Month 12 visit. The rate and 95% confidence interval will be presented by randomization group. All subjects randomized will be included.
Time Frame: 12 month
Population: All randomized subjects are included.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | DBS-f on | DBS-f Off
Number analyzed (Participants) | 21 | 21
participants | 0 [0 to 16.1] | 1 [0.1 to 23.8]

3. Secondary Outcome: ADAS-Cog 13
Description: The mean change from baseline (pre-implant) to 12 months will be calculated in each treatment group. The differences between randomized groups in mean change will be calculated, along with corresponding 2-sided, 95% confidence intervals.
  Instrument is Alzheimer's Disease Assessment Scale - Cognitive subscale. Scores range from 0 to 85 with higher scores meaning worse outcome.
Time Frame: Baseline and 12 months
Population: All randomized subjects
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | DBS-f on | DBS-f Off
Number analyzed (Participants) | 21 | 21
score on a scale | 8.0 (2.2) | 8.0 (1.9)

4. Secondary Outcome: CDR-SB
Description: The mean change from baseline (pre-implant) to 12 months will be calculated in each treatment group. The differences between randomized groups in mean change will be calculated, along with corresponding 2-sided, 95% confidence intervals.
  The scale used is the Clinical Dementia Rating Scale and the score used is the sum of boxes. The scores for this measure range from 0 to 18 with a higher score indicating a worse outcome.
Time Frame: Baseline and 12 months
Population: All randomized subjects with available data. Two subjects in the ON group had missing CDR at 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | DBS-f on | DBS-f Off
Number analyzed (Participants) | 19 | 21
score on a scale | 2.5 (0.4) | 2.6 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent until study exit for each subject. Maximum duration was 48 months.
Description: An independent Clinical Events Committee (CEC) reviewed all reported adverse events. The CEC was responsible for conducting a review of all adverse events reported for study subjects. The CEC will adjudicate and classify all events for relatedness to the study system, study procedure and study requirements. The CEC will determine if any serious device-related adverse event is an unanticipated adverse device effect (UADE).
Arm/Group | DBS-f on | DBS-f Off
All-Cause Mortality (participants affected / at risk) | 1/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 8/21 | 8/21
Other Adverse Events (participants affected / at risk) | 19/21 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBS-f on (N=21) | DBS-f Off (N=21)
UTI (Infections and infestations) | 0 (0) | 1 (1) — Urinary tract infection
Headache (General disorders) | 1 (1) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (4)
Altered mental status (Nervous system disorders) | 1 (1) | 1 (1)
Fall (Nervous system disorders) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) — suspected aortic valve endocarditis
Increased rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
myocardial infarction with stent (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Device infection (Infections and infestations) | 2 (3) | 1 (1)
Abnormal MRI (Surgical and medical procedures) | 0 (0) | 1 (1)
Subdural hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) — bilateral subacute and chronic
Lead misplacement (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBS-f on (N=21) | DBS-f Off (N=21)
Agitation (Nervous system disorders) | 2 (2) | 2 (4)
Anxiety (Nervous system disorders) | 2 (2) | 2 (6)
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Change in Mental Status (Psychiatric disorders) | 1 (1) | 1 (1)
Respiratory Infection (Infections and infestations) | 5 (9) | 4 (6)
Confusion (Nervous system disorders) | 3 (3) | 6 (7)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Delerium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 6 (6) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dizziness (General disorders) | 1 (1) | 2 (2)
Epistaxis (General disorders) | 3 (3) | 0 (0)
Fall (General disorders) | 2 (2) | 5 (17)
Fatigue (General disorders) | 4 (4) | 4 (4)
Fecal Incontinence (Gastrointestinal disorders) | 1 (1) | 2 (2)
Headache (General disorders) | 6 (7) | 7 (7)
Insomnia (General disorders) | 2 (2) | 4 (4)
Irritability (Nervous system disorders) | 2 (2) | 1 (1)
Lethargy (General disorders) | 0 (0) | 2 (2)
Migraine (General disorders) | 2 (3) | 0 (0)
Nausea (General disorders) | 4 (4) | 4 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Paranoid Ideation (Psychiatric disorders) | 1 (3) | 1 (1)
Seizure (Nervous system disorders) | 2 (6) | 0 (0)
Shortness of Breath (General disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary Incontenance (Renal and urinary disorders) | 0 (0) | 2 (2)
visual Hallucinations (Psychiatric disorders) | 1 (1) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
While this feasibility trial was randomized it was not designed with formal hypotheses nor was it powered for analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No